CLINICAL TRIAL: NCT02380534
Title: Use of H.E.L.P. Apheresis in Patients With High Cardiovascular Disease Lp(a)-Related
Brief Title: Use of Apheretic Technologies in Cardiovascular Disease
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding missing
Sponsor: University of Pavia (Other)
Collaborators: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Giuseppe Derosa, MD, PhD, University of Pavia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P-20140023880
Record Dates: First submitted 2015-02-23; First posted 2015-03-05 (Estimated); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Dyslipidemia
Keywords: High level of Lp(a)
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- active procedure (Experimental): High cardiovascular risk patients will undergo H.E.L.P. apheresis.
  Interventions: Procedure: H.E.L.P. apheresis

INTERVENTIONS:
Procedure: H.E.L.P. apheresis — High cardiovascular risk patients will undergo H.E.L.P. apheresis procedure every 3 weeks for 1 year.

SUMMARY:
To evaluate the effects of H.E.L.P. apheresis on lipid profile, Lp(a) level, and some inflammatory adypocytokines in patients with high cardiovascular risk.

ELIGIBILITY:
Inclusion Criteria:

* high Lp(a) not responsive to diet and pharmacological treatment

Exclusion Criteria:

* heart failure
* hepatic failure
* renal failure

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2016-02-04 (Actual)

PRIMARY OUTCOMES:
Lp(a) reduction | 1 year
  We will evaluate the efficacy of apheretic technique through the reduction of Lp(a) in the plasma sample expressed by mg/dL.

SECONDARY OUTCOMES:
Inflammatory adypocytokines | 1 year
  We will evaluate the efficacy of apheretic technique through the improvement of inflammatory adypocytokines in the plasma sample.

OTHER OUTCOMES:
Lipid profile | 1 year
  We will evaluate the efficacy of apheretic technique through the reduction of total cholesterol, LDL and HDL cholesterol, and triglycerides in the plasma sample expressed by mg/dL.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Policlinico S. Matteo, Pavia, Italy